CLINICAL TRIAL: NCT00853788
Title: Genomic and Histological Analysis of Skin Biopsy Specimens as Biomarkers of Systemic Sclerosis and Response to Mycophenolate Mofetil
Brief Title: Skin Biopsy Specimens as Biomarkers of Systemic Sclerosis and Response to Mycophenolate Mofetil
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Monique Hinchcliff, Monique Hinchcliff, MD, MS, Northwestern University
Other Study IDs: STU00004428; 5K12HD055884-02 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; biomarkers; microarray
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin biopsy samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess whether skin biopsy specimens from patients with diffuse cutaneous systemic sclerosis (dcSSc) can be used as biomarkers (measures of activity and type) of disease to predict response to various experimental treatments. There are various experimental treatments being used in the treatment of slceroderma, but there is no way to predict response to any given therapy. The investigators will use DNA microarray to analyze the changes in gene expression in skin biopsies in response to various treatments. Our hypothesis is that the investigators will see changes in gene expression in response to various treatments that will give us insight into the cause of scleroderma. The investigators predict that they will be able to use this information to predict which experimental treatments will be beneficial to individual patients

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is an autoimmune connective tissue disease primarily affecting young to middle-aged women. The pathogenesis of SSc is complex involving interplay of three seemingly diverse processes: autoimmunity, vasculopathy, and fibrosis. Patients experience varying degrees of disabling skin thickening and potentially life-threatening internal organ fibrosis and vasculopathy, but there is no way to accurately predict disease subtype and risk for severity and progression. Current experimental treatments for SSc include oral and intravenous cyclophosphamide and mycophenolate mofetil that blunt the immune response, autologous stem cell transplant that may reset the immune system, and imatinib mesylate that may reduce fibrosis.

Recent exciting genomics research from our lab and our collaborator suggests that skin biopsy samples obtained from patients with SSc have robust alterations in gene expression profiles compared to controls. Changes in expression of genes known to be involved in profibrotic pathways were prominent. The present proposal describes novel experiments to evaluate genomic approaches coupled with clinical data to identify patient subsets, predict response to treatment, and to better understand the molecular basis for disease pathogenesis, and treatment response.

The Northwestern Scleroderma Program (NSP) is a novel multidisciplinary program to accelerate SSc research and provide comprehensive care to >400 SSc patients. Standardized clinical information including demographic, laboratory, and diagnostic data (echocardiography, high resolution chest computerized tomography, and pulmonary function testing) as well as DNA is currently collected on all patients and entered into a clinical database. NSP patients will be offered the option to donate dermal tissue for genomic analysis using a previously established, optimized approach to extract RNA from tissue samples.

We hypothesize that our DNA microarray technique will permit analysis of changes in gene expression from the skin of patients undergoing dermal biopsies before and after treatment and will identify unrecognized profibrotic pathways in addition to providing new, important information regarding known fibrotic pathways. The knowledge gained will not only deepen our understanding of the molecular pathways involved in fibrosis, but also provide a means to reliably predict which patients are likely to respond to various treatments.

Relevance:

SSc is a devastating orphan connective tissue disease with no known cure. There are no disease biomarkers that can accurately predict disease subtype or risk for internal organ involvement and progression at present. Using well-established genomic techniques, the current proposal will investigate if changes in gene expression of profibrotic pathways in dermal biopsies before and after various treatments correlates with clinical response. If so, genonic analysis of dermal tissue may be useful to better understand the molecular pathogenesis of SSc and as a disease biomarker.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* systemic sclerosis

Exclusion Criteria:

* pregnant
* bleeding disorder
* history of delayed wound healing

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diffuse cutaneous systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Hinchcliff, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Faculty Foundation, Chicago, Illinois, United States